CLINICAL TRIAL: NCT03167021
Title: Survey on the Place of Community Pharmacists in the Detection of Cannabis Use: a Student's Point of View
Acronym: CANNACY
Status: Completed | Type: Observational
Sponsor: University Hospital, Clermont-Ferrand (Other)
Responsible Party: Sponsor
Other Study IDs: CHU-333; 2017-A00328-45 (Other: 2017-A00328-45)
Record Dates: First submitted 2017-05-11; First posted 2017-05-25 (Actual); Last update posted 2017-07-07 (Actual); Status verified 2017-05

CONDITIONS: Cannabis Use
Keywords: Cannabis; Community pharmacy; Prevention; Students
MeSH Terms: conditions — Marijuana Abuse | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Students: Students of the Auvergne Rhone Alpes region will be contacted by email thanks to the student associations and scholarity departments. Answer to the survey will be done online.
  Interventions: Other: Survey

INTERVENTIONS:
Other: Survey — This observational and transversal study will be conducted as a survey using the REDCap software and the response to this survey will be done online, in real time, with an automatic, secure and centralized data collection (CHU Clermont-Ferrand).

SUMMARY:
The objective of this survey will be to evaluate the perception by the students (except for medical students, pharmacies) of community pharmacists concerning the management of cannabis consumption. We want to see if the student population perceives the pharmacist as the public health actor of choice, and if they would more easily turn to him or to another health professional (doctor, nurse) in case they need. Discussing possible problematic consumption or for a simple search for information. It will be assessed whether the pharmacist seems to be a good candidate and an element of choice when young adults want to take an intelligence approach to cannabis consumption.

DETAILED DESCRIPTION:
This observational and transversal study will be conducted as a survey using the REDCap software and the response to this survey will be done online, in real time, with an automatic, secure and centralized data collection (CHU Clermont-Ferrand).

Students of the Auvergne Rhone Alpes region will be contacted by email thanks to the student associations and scholarity departments. Answer to the survey will be done online via the following link https://redcap.chu-clermontferrand.fr/surveys/?s=JMRF9FLRJP.

ELIGIBILITY:
Inclusion Criteria:

- Student following a university path in the Auvergne Rhone Alpes region

Exclusion Criteria:

* Medical student
* Pharmacy student
* age < 18-year
* Other than student

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The young and student populations are particularly affected by the use of addictive substances, including alcohol, tobacco and cannabis. Students of the Auvergne Rhone Alpes region will be contacted by email thanks to the student associations and scolarity departments. Answer to the survey will be done online.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Actual)
Dates: Start 2017-04-05 (Actual); Primary Completion 2017-06-02 (Actual); Study Completion 2017-06-02 (Actual)

PRIMARY OUTCOMES:
Role of health professionals in the prevention of cannabis addiction | at day 1
  Students' perceptions (visual analogic scale) of the role of three types of health professionals (community pharmacists, general practitioners and academic health services) in the prevention of cannabis addiction

SECONDARY OUTCOMES:
Role of health professionals for the therapeutic management of cannabis addiction | at day 1
  Assessment of students' perceptions (visual analogic scale) of the role of three types of health professionals (community pharmacists, general practitioners and academic health services) for the therapeutic management of cannabis addiction.
Cannabis consumption | at day 1
  yes/no
Type of cannabis used | at day 1
  marijuana/haschich
Frequency of cannabis use | at day 1
Sought effects of cannabis use | at day 1
  Recreational / Stone / Therapeutic / Other expected effect
Level of knowledge on cannabis | at day 1
  Yes I know the risk / No I don't know the risk
Consumption of cigarettes | at day 1
  yes/no
Consumption of e-cigarettes | at day 1
  yes/no
Consumption of alcohol | at day 1
  yes/no

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Clermont-Ferrand, Clermont-Ferrand, Auvergne, France